CLINICAL TRIAL: NCT00027807
Title: Treatment of Stage IV Breast Cancer With OKT3 x Herceptin Armed Activated T Cells, Low Dose IL-2, And GM-CSF (Phase I Only as of 4-22-09 as Per IRB Approval Date)
Brief Title: Biological Therapy in Treating Women With Stage IV Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Lawrence Lum, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000069072; P30CA022453 (NIH); 2006-130 (Other: Karmanos Cancer Institute); RWMC-0635146; WSU-010307M1F (Other: Wayne State University - Human Investigation Committee); WSU-0312004412 (Other: Wayne State University - Human Investigation Committee)
Record Dates: First submitted 2001-12-07; First posted 2003-01-27 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer; ductal breast carcinoma
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Ductal, Breast | interventions — aldesleukin; Interleukin-2; sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor; Colony-Stimulating Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aldesleukin, Sargramostim & therapeutic autologous lymphocytes (Experimental): Peripheral blood mononuclear cells (PBMC) for the generation of ATC will be collected using 1 or 2 phereses to obtain 8-20 × 109 PBMC for T cell expansion. The PBMC will be activated with OKT3 and expanded in IL-2 to generate from 20-320 ×109 ATC during a maximum of 14 days of culture. Three patients will be treated at each dose level. The dose levels for each infusion are: 5, 10, 20, and 40 billion. Each patient will receive a total of 8 doses of armed ATC given twice weekly for 4 weeks. If the patients encounter toxicities related to armed ATC, the dose and administration will be modified as delineated per the protocol. The patients will also receive subcutaneous injections of IL-2 (3.0 × 105 IU/m2/day) starting 3 days before the 1st armed ATC infusion and ending 7 days after the last armed ATC infusion. GM-CSF (250μg/m2 twice per week) will given subcutaneously to start 3 days before the 1st armed ATC infusion and ending 7 days after the last dose of armed ATC.
  Interventions: Biological: Aldesleukin; Biological: Sargramostim; Biological: therapeutic autologous lymphocytes

INTERVENTIONS:
Biological: Aldesleukin — Subcutaneous injections of IL-2 (3.0 × 105 IU/m2/day) starting 3 days before the 1st armed ATC infusion and ending 7 days after the last armed ATC infusion.
  Other Names: Proleukin ®; IL-2
Biological: Sargramostim — GM-CSF Injections will be given SQ GM-CSF (250 μg/m2/twice weekly), to start 3 days before the first ATC infusion and ending 1 week after the last ATC infusion.
  Other Names: LeukineTM; GM-CSF; Granulocyte-Macrophage Colony Stimulating Factor
Biological: therapeutic autologous lymphocytes — The time for armed-ATC infusions will vary from patient to patient, but the dose of armed-ATC (up to 40 billion) will be given over 30 min.

SUMMARY:
RATIONALE: Biological therapies use different ways to stimulate the immune system and stop cancer cells from growing. Combining different types of biological therapies may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of combining different biological therapies in treating women who have stage IV breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of armed activated T cells given in combination with interleukin-2 and sargramostim (GM-CSF) in women with stage IV breast cancer.
* Determine the toxicity profile of this regimen in these patients.
* Determine the clinical response and overall and progression-free survival of patients treated with this regimen.

OUTLINE: This is a dose-escalation study of armed activated T cells.

Patients undergo peripheral blood mononuclear cell (PBMC) collection. The PBMCs are treated ex vivo with monoclonal antibody OKT3 to form armed activated T cells (ATC). The armed ATC are expanded for 14 days in interleukin-2 (IL-2).

Patients receive armed ATC IV over 30 minutes twice weekly for 4 weeks. Patients also receive IL-2 subcutaneously (SC) once daily and sargramostim (GM-CSF) SC twice weekly beginning 3 days before the first infusion of armed ATC and continuing until 7 days after the last infusion of armed ATC.

Cohorts of 3-6 patients receive escalating doses of armed ATC until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, additional patients are treated at that dose.

Patients are followed at 1, 2, and 5 months and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 15-30 patients will be accrued for the phase I portion of this study and a total of 18-33 patients will be accrued for the phase II portion of this study within 4-6 years.

PLEASE NOTE: THIS STUDY WAS INTENDED TO BE A PHASE I/II STUDY, BUT NEVER MOVED FORWARD TO PHASE II. (4-22-09)

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Phase I:

* Histologically confirmed infiltrating ductal carcinoma of the breast
* Metastatic disease

  * Clinically asymptomatic with non-life-threatening metastases allowed
* Measurable or evaluable disease by radiograph, CT scan, MRI, nuclear medicine bone scan, or physical examination

  * No measurable disease allowed if tumor or metastasis has been removed or successfully treated prior to study
* No rapidly progressive symptomatic disease affecting major organ systems (e.g., lungs and liver)
* Stable or unstable disease for 3 months on hormonal therapy
* Stable or unstable disease for at least 1 month after chemotherapy
* No active brain metastases

  * Brain metastases previously treated with definitive radiotherapy and/or surgical resection allowed
* Hormone receptor status:

  * Estrogen and progesterone receptor status known

Phase II:

* All Phase I criteria
* HER2/neu overexpression (2+ or 3+) by immunohistochemistry

  * Prior trastuzumab (Herceptin) allowed if disease still overexpresses HER2/neu

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* Karnofsky 70-100% OR
* ECOG 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* Granulocyte count at least 1,500/mm^3
* Platelet count at least 50,000/mm^3
* Hemoglobin at least 8 g/dL

Hepatic:

* Bilirubin less than 1.5 times normal
* SGOT less than 1.5 times normal

Renal:

* Creatinine no greater than 1.8 mg/dL
* Creatinine clearance at least 60 mL/min
* BUN no greater than 1.5 times normal

Cardiovascular:

* No myocardial infarction within the past year
* No prior myocardial infarction with coronary symptoms requiring medication and/or depressed left ventricular function (LVEF less than 50% by MUGA)
* No angina or coronary symptoms requiring medication and/or with depressed left ventricular function (LVEF less than 50% by MUGA)
* No congestive heart failure requiring medical management
* LVEF at least 50% at rest by MUGA
* No uncontrolled hypertension (i.e., systolic blood pressure [BP] ≥ 130 mm Hg or diastolic BP ≥ 80 mm Hg)

Pulmonary:

* FEV1, DLCO, and FVC at least 50% predicted

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No other serious medical or psychiatric illness that would preclude study participation
* No other prior or concurrent malignancy within the past 5 years except curatively treated squamous cell carcinoma in situ of the cervix, basal cell skin cancer, or any other curatively treated disease in complete remission

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* Prior trastuzumab allowed for phase I

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy

Endocrine therapy:

* See Disease Characteristics
* Concurrent hormonal therapy for breast cancer must continue during study
* No other concurrent hormonal therapy except steroids for adrenal failure, septic shock, or pulmonary toxicity or hormonal therapy for non-disease-related conditions (e.g., insulin for diabetes)

Radiotherapy:

* See Disease Characteristics

Surgery:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2001-10; Primary Completion 2010-09 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | The dose at which dose-limiting toxicity occurs is defined as that dose at which 2 or more of 6 patients at that dose level have their infusions stopped due to toxicities or receive less than 80% of the planned dose.
Toxicity profile | Months 1, 2, 5 and 11, then every 6 months
Clinical responses | Months: 1, 2, 5 and 11, then every 6 months
Overall survival and progression-free survival | The interval from the beginning of immunotherapy to the time of death or for progression free survival it is defined as the interval from the beginning of immunotherapy to progression

SECONDARY OUTCOMES:
Immune changes | 1 (+ 7 days), 2 (+ 7 days), 5 months (+ 7 days), then every 6months (+ 7 days) (immune evaluations will also be performed after the 4th and 8th infusion of Her2Bi armed ATC and within 1week of the completion of HER2Bi armed ATC)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence G. Lum, MD, DSc, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

REFERENCES:
- [Background] Lum LG, Rathore R, Colvin GA, et al.: Targeting HER2/neu tumor cells with anti-CD3 activated T cells: clinical trials and trafficking studies. [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-719, 2003.
- [Result] Grabert RC, Smith JA, Tiggs JC, et al.: Anti-CD3 activated T cells (ATC) armed with OKT3 x Herceptin Bispecific antibody (Her2Bi), survive and divide, and secrete cytokines and chemokines after multiple cycles of killing directed at Her2/neu+ (Her2) tumor targets. [Abstract] Proceedings of the 94th Annual Meeting of the American Association of Cancer Research 44: A-2872, 565, 2003.
- [Result] Sen M, Wankowski DM, Garlie NK, Siebenlist RE, Van Epps D, LeFever AV, Lum LG. Use of anti-CD3 x anti-HER2/neu bispecific antibody for redirecting cytotoxicity of activated T cells toward HER2/neu+ tumors. J Hematother Stem Cell Res. 2001 Apr;10(2):247-60. doi: 10.1089/15258160151134944. PMID 11359672
- [Result] Lum LG, Thakur A, Al-Kadhimi Z, Colvin GA, Cummings FJ, Legare RD, Dizon DS, Kouttab N, Maizel A, Colaiace W, Liu Q, Rathore R. Targeted T-cell Therapy in Stage IV Breast Cancer: A Phase I Clinical Trial. Clin Cancer Res. 2015 May 15;21(10):2305-14. doi: 10.1158/1078-0432.CCR-14-2280. Epub 2015 Feb 16. PMID 25688159
- [Derived] Park JA, Santich BH, Xu H, Lum LG, Cheung NV. Potent ex vivo armed T cells using recombinant bispecific antibodies for adoptive immunotherapy with reduced cytokine release. J Immunother Cancer. 2021 May;9(5):e002222. doi: 10.1136/jitc-2020-002222. PMID 33986124